CLINICAL TRIAL: NCT01383603
Title: Identification of Potential Biomarkers of Peptide Immunotherapy. Part 2 - Gene Array Analysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES-004
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Cat Allergy
Keywords: Cat Allergy; Rhinoconjunctivitis; Immunotherapy; Cat-PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cat-PAD (Experimental)
  Interventions: Biological: Cat-PAD

INTERVENTIONS:
Biological: Cat-PAD — Intradermal injection 1 x 4 administrations 4 weeks apart

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis. Cat-PAD is a novel, synthetic, allergen derived peptide desensitising vaccine currently being developed for treatment of cat allergy.

At present, the efficacy of immunotherapy (peptide or otherwise) can only be established at the conclusion of therapy. No reliable predictive biomarkers of clinical efficacy currently exist. Identification of surrogate biomarkers of clinical efficacy, would facilitate clinical development of peptide immunotherapy vaccines, in addition to providing an improved understanding of the underlying molecular mechanisms of efficacy, thus providing new leads for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Weight >50 kg.
* A minimum 1-year documented history of rhinoconjunctivitis on exposure to cats.
* Positive skin prick test to cat allergen.
* Subjects must have regular exposure to a cat in their normal living or working circumstances throughout the course of the study.
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion Criteria:

* History of asthma
* History of anaphylaxis to cat allergen
* History of allergen immunotherapy in the previous 10 years, or in the previous 3 years for pre-seasonal immunotherapy treatments
* History of any significant disease or disorder (e.g. autoimmune, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment, severe atopic dermatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Identification of a change in gene expression over the course of and potentially attributable to Cat-PAD treatment. | 6 months following treatment

SECONDARY OUTCOMES:
Symptom scores for ocular and nasal symptoms | 4 weeks following treatment
Interleukin production and eosinophil level changes | 4 weeks following treatment
Functional genomic changes | 4 weeks following treatment
Changes in urine metabolomic profiles | 4 weeks following treatment

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Neighbour H, Soliman M, Steacy LM, Hickey P, Forbes B, Larche M, Ellis AK. The Allergic Rhinitis Clinical Investigator Collaborative (AR-CIC): verification of nasal allergen challenge procedures in a study utilizing an investigational immunotherapy for cat allergy. Clin Transl Allergy. 2018 Apr 12;8:15. doi: 10.1186/s13601-018-0198-7. eCollection 2018. PMID 29682277